CLINICAL TRIAL: NCT01880164
Title: Cost Effectiveness of Nonoperative Management for Adult Spinal Deformity Associated With Low Grade Scoliosis: A Prospective Pilot Study to Evaluate Disease Burden and Longitudinal Study Feasibility
Brief Title: Cost Effectiveness of Nonoperative Management for Adult Spinal Deformity
Acronym: HEO
Status: Completed | Type: Observational
Sponsor: Shay Bess (Other)
Collaborators: DePuy Spine (Industry); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Shay Bess, President, ISSGF, International Spine Study Group Foundation
Organization: International Spine Study Group Foundation (Other)
Other Study IDs: 2108
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Spinal Deformity
Keywords: Scoliosis; Kyphosis; Sagittal plane deformity
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nonoperative: Adult spinal deformity (degenerative or idiopathic) with an ODI of 30 or greater

SUMMARY:
Quantify the efficacy and cost of nonoperative treatment modalities used for adult spinal deformity.

DETAILED DESCRIPTION:
1. Identify disease burden associated with adult spinal deformity (ASD) using quality adjusted life year (QALY) analysis.
2. Identify disease burden of specific demographic and radiographic features associated with ASD.
3. Compare disease burden of ASD to other musculoskeletal and non-musculoskeletal diseases.
4. Identify efficacy of specific nonoperative treatment modalities to treat ASD and identify specific clinical and radiographic features of ASD responsive to nonoperative treatment modalities.
5. Compare QALY and ICER values for different ASD nonoperative treatment modalities to previously established QALY and ICER for values for operative and nonoperative treatment modalities for degenerative hip and knee disease, coronary artery disease, insulin dependent diabetes, and hypertension.
6. Evaluate the cost and work hours associated with data collection and minimum 85% patient follow up.
7. Evaluate patient characteristics associated with poor patient compliance for study follow up including demographic, radiographic and HRQOL values and for reasons for cross-over to operative treatment for ASD.
8. Establish standardized data collection methodology for economic based outcome studies based upon patient demographics and HRQOL values.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years of age at the time of enrollment.
2. ODI ≥30
3. Adult degenerative or idiopathic lumbar scoliosis 10-40° as measured by the Cobb angle technique
4. Sagittal plane deformity by SRS Schwab classification with at least one modifier ++ or two modifiers + and associated coronal cobb of at least 10 degrees

Exclusion Criteria:

1. Adult degenerative or idiopathic scoliosis with a curvature of the spine measuring <10 degrees or >40 degrees
2. Diagnosis of scoliosis other than degenerative or idiopathic (i.e. neuromuscular, congenital, etc.)
3. Cardiopulmonary disease or comorbidities that preclude surgical intervention
4. Patient not deemed surgical candidate by treating surgeon
5. Patient unwilling to commit to monthly phone interviews or completion of necessary questionnaires or inability to return for defined follow up time points. Patients unwilling to comply with study protocol will not be offered enrollment into the study, regardless of meeting inclusion criteria.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult spinal deformity patients
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Initial visit and six months post enrollment
  This questionnaire has been designed to provide information as to how back pain affects ability to manage in everyday life. Score must be equal to or greater than 30 for eligibility to enroll.

SECONDARY OUTCOMES:
Radiographs | Initial visit (Day 1)
  Coronal and sagittal radiographic views of the spine obtained to assess coronal curvature and sagittal balance.

OTHER OUTCOMES:
SRS22r | Initial (Day1) and six months post enrollment
  Assess pain, function, self image, and mental health.
EQ5D-3L | Initial (Day1) and six months post enrollment
  Assess health state (best imaginable vs worst imaginable).
Work Productivity and Activity Impairment (WPAI:SHP) | Initial (Day1) and six months post enrollment
  Assess ability to work and perform regular activities as relates to spinal deformity.
NRS | Initial (Day1) and six months post enrollment
  Assess back and leg pain.
Resource Utilization (RRU) | Initial clinic visit (Day1) , Phone interviews at 1, 2, 3, 4, and 5 months, and 6 months clinic visit
  Document nonoperative treatment modalities, such as observation only, pain medicine, physical therapy, chiropractic care, injections, diagnostic radiology, emergency visits, and other therapies. Analysis of this data will determine cost associated with nonoperative care for adult spinal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Shay Bess, MD, Principal Investigator — Rocky Mountain Scoliosis and Spine
Locations (10):
- United States (10):
  - University of California - Davis, Sacramento, California
  - University of California - San Francisco Medical Center, San Francisco, California
  - Rocky Mountain Scoliosis and Spine, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Washington University at St. Louis, St Louis, Missouri
  - NYU Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avorn J. Debate about funding comparative-effectiveness research. N Engl J Med. 2009 May 7;360(19):1927-9. doi: 10.1056/NEJMp0902427. No abstract available. PMID 19420361
- [Background] Baldus C, Bridwell KH, Harrast J, Edwards C 2nd, Glassman S, Horton W, Lenke LG, Lowe T, Mardjetko S, Ondra S, Schwab F, Shaffrey C. Age-gender matched comparison of SRS instrument scores between adult deformity and normal adults: are all SRS domains disease specific? Spine (Phila Pa 1976). 2008 Sep 15;33(20):2214-8. doi: 10.1097/BRS.0b013e31817c0466. PMID 18794764
- [Background] Berven S, Deviren V, Demir-Deviren S, Hu SS, Bradford DS. Studies in the modified Scoliosis Research Society Outcomes Instrument in adults: validation, reliability, and discriminatory capacity. Spine (Phila Pa 1976). 2003 Sep 15;28(18):2164-9; discussion 2169. doi: 10.1097/01.BRS.0000084666.53553.D6. PMID 14501930
- [Background] Bonham AC, Rich EC, Davis DA, Longnecker DE, Heinig SJ. Commentary: Putting evidence to work: an expanded research agenda for academic medicine in the era of health care reform. Acad Med. 2010 Oct;85(10):1551-3. doi: 10.1097/ACM.0b013e3181effdbc. PMID 20703148
- [Background] Bridwell KH, Berven S, Glassman S, Hamill C, Horton WC 3rd, Lenke LG, Schwab F, Baldus C, Shainline M. Is the SRS-22 instrument responsive to change in adult scoliosis patients having primary spinal deformity surgery? Spine (Phila Pa 1976). 2007 Sep 15;32(20):2220-5. doi: 10.1097/BRS.0b013e31814cf120. PMID 17873814
- [Background] Bridwell KH, Glassman S, Horton W, Shaffrey C, Schwab F, Zebala LP, Lenke LG, Hilton JF, Shainline M, Baldus C, Wootten D. Does treatment (nonoperative and operative) improve the two-year quality of life in patients with adult symptomatic lumbar scoliosis: a prospective multicenter evidence-based medicine study. Spine (Phila Pa 1976). 2009 Sep 15;34(20):2171-8. doi: 10.1097/BRS.0b013e3181a8fdc8. PMID 19752703
- [Background] Carter OD, Haynes SG. Prevalence rates for scoliosis in US adults: results from the first National Health and Nutrition Examination Survey. Int J Epidemiol. 1987 Dec;16(4):537-44. doi: 10.1093/ije/16.4.537. PMID 3501989
- [Background] Deyo RA, Mirza SK, Martin BI, Kreuter W, Goodman DC, Jarvik JG. Trends, major medical complications, and charges associated with surgery for lumbar spinal stenosis in older adults. JAMA. 2010 Apr 7;303(13):1259-65. doi: 10.1001/jama.2010.338. PMID 20371784
- [Background] Everett CR, Patel RK. A systematic literature review of nonsurgical treatment in adult scoliosis. Spine (Phila Pa 1976). 2007 Sep 1;32(19 Suppl):S130-4. doi: 10.1097/BRS.0b013e318134ea88. PMID 17728680
- [Background] Garber AM, Tunis SR. Does comparative-effectiveness research threaten personalized medicine? N Engl J Med. 2009 May 7;360(19):1925-7. doi: 10.1056/NEJMp0901355. No abstract available. PMID 19420360
- [Background] Garrison KR, Donell S, Ryder J, Shemilt I, Mugford M, Harvey I, Song F. Clinical effectiveness and cost-effectiveness of bone morphogenetic proteins in the non-healing of fractures and spinal fusion: a systematic review. Health Technol Assess. 2007 Aug;11(30):1-150, iii-iv. doi: 10.3310/hta11300. PMID 17669279
- [Background] Glassman SD, Berven S, Kostuik J, Dimar JR, Horton WC, Bridwell K. Nonsurgical resource utilization in adult spinal deformity. Spine (Phila Pa 1976). 2006 Apr 15;31(8):941-7. doi: 10.1097/01.brs.0000209318.32148.8b. PMID 16622386
- [Background] Glassman SD, Bridwell K, Dimar JR, Horton W, Berven S, Schwab F. The impact of positive sagittal balance in adult spinal deformity. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2024-9. doi: 10.1097/01.brs.0000179086.30449.96. PMID 16166889
- [Background] Glassman SD, Carreon LY, Shaffrey CI, Polly DW, Ondra SL, Berven SH, Bridwell KH. The costs and benefits of nonoperative management for adult scoliosis. Spine (Phila Pa 1976). 2010 Mar 1;35(5):578-82. doi: 10.1097/BRS.0b013e3181b0f2f8. PMID 20118843
- [Background] Glassman SD, Polly DW, Dimar JR, Carreon LY. The cost effectiveness of single-level instrumented posterolateral lumbar fusion at 5 years after surgery. Spine (Phila Pa 1976). 2012 Apr 20;37(9):769-74. doi: 10.1097/BRS.0b013e3181e03099. PMID 20489676
- [Background] Hirth RA, Bloom BS, Chernew ME, Fendrick AM. Patient, physician, and payer perceptions and misperceptions of willingness to pay for diagnostic certainty. Int J Technol Assess Health Care. 2000 Winter;16(1):35-49. doi: 10.1017/s0266462300016147. PMID 10815352
- [Background] Hirth RA, Chernew ME, Miller E, Fendrick AM, Weissert WG. Willingness to pay for a quality-adjusted life year: in search of a standard. Med Decis Making. 2000 Jul-Sep;20(3):332-42. doi: 10.1177/0272989X0002000310. PMID 10929856
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Background] Lafage V, Schwab F, Patel A, Hawkinson N, Farcy JP. Pelvic tilt and truncal inclination: two key radiographic parameters in the setting of adults with spinal deformity. Spine (Phila Pa 1976). 2009 Aug 1;34(17):E599-606. doi: 10.1097/BRS.0b013e3181aad219. PMID 19644319
- [Background] Lafage V, Schwab F, Skalli W, Hawkinson N, Gagey PM, Ondra S, Farcy JP. Standing balance and sagittal plane spinal deformity: analysis of spinopelvic and gravity line parameters. Spine (Phila Pa 1976). 2008 Jun 15;33(14):1572-8. doi: 10.1097/BRS.0b013e31817886a2. PMID 18552673
- [Background] Laupacis A, Feeny D, Detsky AS, Tugwell PX. How attractive does a new technology have to be to warrant adoption and utilization? Tentative guidelines for using clinical and economic evaluations. CMAJ. 1992 Feb 15;146(4):473-81. PMID 1306034
- [Background] Loomes G, McKenzie L. The use of QALYs in health care decision making. Soc Sci Med. 1989;28(4):299-308. doi: 10.1016/0277-9536(89)90030-0. PMID 2649989
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] McCabe C, Claxton K, Culyer AJ. The NICE cost-effectiveness threshold: what it is and what that means. Pharmacoeconomics. 2008;26(9):733-44. doi: 10.2165/00019053-200826090-00004. PMID 18767894
- [Background] Perennou D, Marcelli C, Herisson C, Simon L. Adult lumbar scoliosis. Epidemiologic aspects in a low-back pain population. Spine (Phila Pa 1976). 1994 Jan 15;19(2):123-8. doi: 10.1097/00007632-199401001-00001. PMID 8153817
- [Background] Ridyard CH, Hughes DA. Methods for the collection of resource use data within clinical trials: a systematic review of studies funded by the UK Health Technology Assessment program. Value Health. 2010 Dec;13(8):867-72. doi: 10.1111/j.1524-4733.2010.00788.x. Epub 2010 Oct 12. PMID 20946187
- [Background] Rihn JA, Berven S, Allen T, Phillips FM, Currier BL, Glassman SD, Nash DB, Mick C, Crockard A, Albert TJ. Defining value in spine care. Am J Med Qual. 2009 Nov-Dec;24(6 Suppl):4S-14S. doi: 10.1177/1062860609349214. PMID 19890180
- [Background] Russell LB, Gold MR, Siegel JE, Daniels N, Weinstein MC. The role of cost-effectiveness analysis in health and medicine. Panel on Cost-Effectiveness in Health and Medicine. JAMA. 1996 Oct 9;276(14):1172-7. PMID 8827972
- [Background] Schwab F, Dubey A, Gamez L, El Fegoun AB, Hwang K, Pagala M, Farcy JP. Adult scoliosis: prevalence, SF-36, and nutritional parameters in an elderly volunteer population. Spine (Phila Pa 1976). 2005 May 1;30(9):1082-5. doi: 10.1097/01.brs.0000160842.43482.cd. PMID 15864163
- [Background] Schwab F, Lafage V, Patel A, Farcy JP. Sagittal plane considerations and the pelvis in the adult patient. Spine (Phila Pa 1976). 2009 Aug 1;34(17):1828-33. doi: 10.1097/BRS.0b013e3181a13c08. PMID 19644334
- [Background] Smith JS, Shaffrey CI, Berven S, Glassman S, Hamill C, Horton W, Ondra S, Schwab F, Shainline M, Fu KM, Bridwell K; Spinal Deformity Study Group. Operative versus nonoperative treatment of leg pain in adults with scoliosis: a retrospective review of a prospective multicenter database with two-year follow-up. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1693-8. doi: 10.1097/BRS.0b013e3181ac5fcd. PMID 19770610
- [Background] Testa MA, Nackley JF. Methods for quality-of-life studies. Annu Rev Public Health. 1994;15:535-59. doi: 10.1146/annurev.pu.15.050194.002535. PMID 8054098
- [Background] Torrance GW. Measurement of health state utilities for economic appraisal. J Health Econ. 1986 Mar;5(1):1-30. doi: 10.1016/0167-6296(86)90020-2. PMID 10311607
- [Background] Tosteson AN, Lurie JD, Tosteson TD, Skinner JS, Herkowitz H, Albert T, Boden SD, Bridwell K, Longley M, Andersson GB, Blood EA, Grove MR, Weinstein JN; SPORT Investigators. Surgical treatment of spinal stenosis with and without degenerative spondylolisthesis: cost-effectiveness after 2 years. Ann Intern Med. 2008 Dec 16;149(12):845-53. doi: 10.7326/0003-4819-149-12-200812160-00003. PMID 19075203
- [Background] Tosteson AN, Skinner JS, Tosteson TD, Lurie JD, Andersson GB, Berven S, Grove MR, Hanscom B, Blood EA, Weinstein JN. The cost effectiveness of surgical versus nonoperative treatment for lumbar disc herniation over two years: evidence from the Spine Patient Outcomes Research Trial (SPORT). Spine (Phila Pa 1976). 2008 Sep 1;33(19):2108-15. doi: 10.1097/brs.0b013e318182e390. PMID 18777603